CLINICAL TRIAL: NCT02656966
Title: Auricular Acupuncture vs. Standard Therapy for Treatment of Preoperative Anxiety in Patients Scheduled for Ambulatory Gynaecological Surgery - a Pilot Non-randomized Controlled Trial
Brief Title: Auricular Acupuncture for Treatment of Preoperative Anxiety
Acronym: AcuAnx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB 158/15
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular acupuncture + standard therapy (Active Comparator): Patients, who will wish acupuncture, will receive this intervention, in addition to standard therapy
  Interventions: Device: Auricular acupuncture
- Standard therapy alone (No Intervention): Patients who do not wish acupuncture will be asked if they will fill in the study questionnaire

INTERVENTIONS:
Device: Auricular acupuncture — Five ear acupuncture points: MA-IC, MA-TF1, MA-SC, MA-AT1 and MA-TG will be needled bilaterally in patients, who will wish to receive AA. Indwelling fixed "New Pyonex" needles (length: 1.5 mm, diameter: 0.22 mm; Seirin Corp., Shizuoka City, Japan) will be used for AA.
  Arms: Auricular acupuncture + standard therapy

SUMMARY:
In this prospective nonrandomized study the investigators are going to investigate whether auricular acupuncture with indwelling fixed needles is feasible for treatment of preoperative anxiety.

Patients, scheduled for ambulatory gynecologic surgery, will be asked, if they wish to receive auricular acupuncture (AA) against preoperative anxiety. The patients who will not wish AA, will be asked to take part in questioning (State-Trait-Anxiety-Inventory (STAI) questionnaire) and will form the control group. The preoperative anxiety using STAI, as well as the duration and quality of sleep on the night before surgery, the incidence of side effects, blood pressure and heart rate will be the outcome measures in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anaesthesiologists physical status of I to II scheduled for elective ambulatory gynaecological surgery under standardized general anaesthesia
2. Surgery time does not exceed 60 minutes
3. Patients without previous opioid and psychotropic medication
4. Patients aged between 19 and 55 years, able to fill in the STAI questionnaire
5. Patients who have given written informed consent

Exclusion Criteria:

1. Current psychiatric disease
2. Local skin infection at the sites of acupuncture
3. Aged < 19 or > 55 years
4. Failure to follow the standardized schema of general anaesthesia
5. Surgery time more than 60 minutes
6. Intraoperative complications (bleeding, required blood transfusion more than 6 units of packed cells, cardiovascular instability, required catecholamines)
7. Patients who consumed opioid medication at least 6 months before surgery
8. Patients who are unable to understand the consent form or to fill in the STAI questionnaire

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Situational anxiety_1 | Situational anxiety_1 will be measured on the day before surgery before auricular acupuncture
  State (situational) anxiety will be measured using State-Trait-Anxiety Inventory (STAI).
Situational anxiety_2 | Situational anxiety_2 will be measured and in the evening of the day before surgery
  State (situational) anxiety will be measured using State-Trait-Anxiety Inventory
Situational anxiety_3 | Situational anxiety_3 will be measured on the day of surgery immediately before the operation
  State (situational) anxiety will be measured using State-Trait-Anxiety Inventory

SECONDARY OUTCOMES:
Heart rate | On the day of surgery before the surgery
Blood pressure | On the day of surgery before the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wunsch JK, Klausenitz C, Janner H, Hesse T, Mustea A, Hahnenkamp K, Petersmann A, Usichenko TI. Auricular acupuncture for treatment of preoperative anxiety in patients scheduled for ambulatory gynaecological surgery: a prospective controlled investigation with a non-randomised arm. Acupunct Med. 2018 Aug;36(4):222-227. doi: 10.1136/acupmed-2017-011456. Epub 2018 Jul 9. PMID 29986900